CLINICAL TRIAL: NCT01447667
Title: Magnetic Resonance Elastography Score Reflecting Hepatic Fibrosis as an Independent Predictor for Recurrence of Hepatocellular Carcinoma After Radiofrequency Ablation Therapy
Brief Title: Magnetic Resonance Elastography (MRE) as a Predictor of HCC Recurrence After Radiofrequency Ablation (RFA)
Acronym: MRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Clinical professor, M.D., Ph.D., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRE
Record Dates: First submitted 2011-09-26; First posted 2011-10-06 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hepatic Fibrosis; Hepatocellular Carcinoma
Keywords: Hepatic fibrosis; Magnetic resonance elastography; Hepatocellular carcinoma; Recurrence
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic resonance elastography (Experimental): Magnetic resonance elastography before radiofrequency ablation therapy will be performed.
  Interventions: Procedure: Magnetic resonance elastography

INTERVENTIONS:
Procedure: Magnetic resonance elastography — Magnetic resonance elastography before RFA and Liver biopsy of 2 HCC tissue and 2 non tumor liver parenchyma tissue

SUMMARY:
The purpose of this study is to determine:

* The efficacy of MRE score as a predictor of HCC recurrence within 2 years after RFA treatment
* The efficacy of each indicator (MRE score, non-invasive serum markers) compared to the gold-standard histology score predicting hepatic fibrosis

DETAILED DESCRIPTION:
To evaluate whether MRE score reflecting hepatic fibrosis can predict the recurrence of HCC within 2 years after RFA treatment

* Local recurrence/intrahepatic distant recurrence
* Multivariable analysis including several related factors to find whether MRE score is an independent predictor of HCC recurrence even after adjusting other factors (etiology of liver disease, size of HCC, vessel invasion, HBsAg titer, etc.)

To find the efficacy of each indicator (MRE score, non-invasive serum markers) compared to the gold-standard histology score predicting hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as single hypervascular hepatocellular carcinoma initially
* AJCC stage I HCC
* Child-Pugh class A
* Planning radiofrequency ablation for HCC
* Voluntary agreement for this study

Exclusion Criteria:

* Decreased kidney function (GFR < 70 mL/min/kg)
* Contraindication to MRI (pacemaker, defibrillator)
* Contrast media hypersensitivity
* Other primary malignancy
* Acute viral hepatitis
* Prior history of liver transplantation
* Thrombosis in splenic vein or portal vein
* Patients who were enrolled to other clinical trials within 4 weeks
* Other severe chronic disease or psychiatric disease
* Pregnant or milk-feeding women
* Patients with coagulopathy, high risk of bleeding for the liver biopsy
* Patients who disagree to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who experienced HCC recurrence after RFA | within 2 years after RFA procedure
  To see whether MRE score reflecting hepatic fibrosis predicts the recurrence of HCC within 2 years after RFA treatment

SECONDARY OUTCOMES:
Sensitivity and specificity of each indicator of hepatic fibrosis compared to the gold-standard histology score | 2 years after RFA
  To find efficacy of each indicator (MRE, noninvasive serum markers such as APRI, P2/MS) compared to the gold-standard histology score in predicting hepatic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No